CLINICAL TRIAL: NCT05502744
Title: Emergency Versus Elective Cholecystectomy in Acute Cholecystitis in the Era of Laparoscopy: A Prospective Randomized Comparative Study
Brief Title: Emergency Versus Elective Cholecystectomy in Acute Cholecystitis in the Era of Laparoscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karam Ezz Rabie, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Still not known
Record Dates: First submitted 2022-08-06; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Versus Elective Cholecystectomy in Acute Cholecystitis in the Era of Laparoscopy (Experimental): A Prospective Randomized Comparative Study.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy is the standard treatment for acute cholecystitis due to the advantages of small wounds, less use of abdominal drains , less need for antibiotics and analgesics and less postoperative hospital stay time.Laparoscopic cholecystectomy in acute cholecystitis may be performed as soon as begging of the symptoms called emergency or urgent and maybe scheduled in advance after controlling acute attack after 6-8weeks called elective.
  Other Names: Emergency versus elective cholecystectomy in acute cholecystits in the era of laproscopy

SUMMARY:
The aim of study is compare outcome of patients undergoing early laparoscopic cholecystectomy within 72 hours from the begging of symptoms to those of patients managed conservatively and operated late after 6-8weeks after the inflammatory reaction has subsided.

DETAILED DESCRIPTION:
Acute cholecystitis is considered one of the most common acute surgical problems. It includes typical symptoms of pain in right hypochondrium, fever, increased leucocytes count and abdominal US used to confirm this clinical diagnosis. Laparoscopic cholecystectomy (LC) is the standard treatment for acute cholecystitis due to the advantages of small wounds, less use of abdominal drains , less need for antibiotics and analgesics and less postoperative hospital stay time.Laparoscopic cholecystectomy in acute cholecystitis may be performed as soon as begging of the symptoms called emergency or urgent laparoscopic cholecystectomy and maybe scheduled in advance after controlling acute attack after 6-8weeks called elective laparoscopic cholecystectomy . Emergency laparoscopic cholecystectomy has advantage of a decreased hospital stay and avoids the risk of emergency admission for non-resolved or recurrent symptoms, which is associated with an increase in morbidity, pain and delayed return to work. Also, some trials showed increased morbidity with elective laparoscopic cholecystectomy mostly due to biliary disease while patients await surgery. Comparative studies are deficient in evaluation of outcomes of emergency cholecystectomy and elective cholecystectomy in acute cholecystitis. So the interest of our study is to compare between the emergency laparoscopic cholecystectomy and elective laparoscopic cholecystectomy regarding the feasibility and the safety of the first.

ELIGIBILITY:
Inclusion Criteria:

1. age less than 70 years.
2. fit for surgery.

Exclusion Criteria:

1. patients with co-existent common bile duct stones based on imaging and biochemical criteria.
2. Patients with Pancreatitis .
3. Patients with previous upper abdominal surgery.
4. Significant medical disease rendering patient unfit for Laparoscopic surgery (e.g.Chronic Pulmonary Disease, significant Cardiac Disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-14 (Estimated); Primary Completion 2022-09-14 (Estimated); Study Completion 2023-08-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative complications in urgent versus elective lap cholecystostomy. | Intraoperative time
  Collect results and see.

SECONDARY OUTCOMES:
Incidence of postoperative complications in urgent versus elective lap cholecystectomy. | 6 months.
  Collect results and see.